CLINICAL TRIAL: NCT03900533
Title: Emotion Regulation Group Skills Training for Adolescents and Parents: A Randomized Controlled Study in a Clinical Setting
Brief Title: Emotion Regulation Group Skills Training for Adolescents and Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Maria Zetterqvist, Principal Investigator, Region Östergötland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/264-31
Record Dates: First submitted 2019-03-29; First posted 2019-04-03 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Behavioral Symptoms; Emotional Instability
Keywords: child psychiatry; emotion regulation skills training
MeSH Terms: conditions — Behavioral Symptoms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjunctive group emotion regulation skills training (Experimental): Participants will receive a 7 week group emotion regulation skills training together with parents adjacent to treatment as usual provided by the child- and adolescent psychiatric clinic
  Interventions: Behavioral: Adjunctive group emotion regulation skills training
- Treatment as usual (TAU) (Active Comparator): Participants will receive treatment as usual for 7 weeks as provided by the child- and adolescent psychiatric clinic
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Adjunctive group emotion regulation skills training — The adjunctive emotion regulation skills training is delivered in a group format once a week during 7 weeks to adolescents and parents jointly together with treatment as usual
  Arms: Adjunctive group emotion regulation skills training
Behavioral: Treatment as usual — Treatment as usual at the child- and adolescent psychiatric clinic is delivered during 7 weeks
  Arms: Treatment as usual (TAU)

SUMMARY:
To evaluate if emotion regulation group therapy skills training for adolescents and parents is an efficacious treatment when delivered as adjunctive to treatment as usual compared to a control group consisting of treatment as usual.

ELIGIBILITY:
Inclusion criteria:

* Being enrolled as a patient at the child- and adolescent psychiatric clinic in Linköping
* Having an adult participant joining the skills training
* Being between the ages of 14-17 years
* Having sufficient knowledge of the Swedish language

Exclusion criteria:

* Clinical diagnosis of schizophrenia
* Clinical diagnosis of psychosis
* Clinical diagnosis of severe anorexia nervosa
* Clinical diagnosis of severe autism spectrum disorder
* Having a cognitive disability
* Having an ongoing drug or alcohol abuse
* Clinical diagnosis of bipolar disorder
* Insufficient knowledge of the Swedish language

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Difficulties with Emotion Regulation Scale (DERS) | Change from baseline at 7 weeks and at 3 months
  Difficulties with Emotion Regulation Scale measures difficulties with emotion regulation. It contains a total of 36 items that are rated on a Likert scale between 1-5. Total score ranges between 36-180 with higher scores indicating more difficulties with emotion regulation. The scale has 6 subscales: nonacceptance (ranging from 6-30); goals (ranging from 5-25); impulse (ranging from 6-30); awareness (ranging from 6-30); strategies (ranging from 8-40) and clarity (ranging from 5-25).

SECONDARY OUTCOMES:
Beck's Anxiety Inventory (BAI) | Change from baseline at 7 weeks and at 3 months
  Beck's Anxiety Inventory measures symptoms of anxiety with 21 items rated on a four-graded scale (0-3). Total scores range from 0-63. Higher scores indicate higher levels of anxiety.
Montgomery Åsberg Depression Rating Scale, self-report version (MADRS-S). | Change from baseline at 7 weeks and at 3 months
  Montgomery Åsberg Depression Rating Scale measures symptoms of depression. Its main purpose is to monitor the development of symptoms during treatment. The scale consists of 9 items, which are graded from zero to six. Total scores range from 0-54. Higher scores indicate higher level of depression symptoms.
Global Assessment Scale for Children (C-GAS) | Change from baseline at 7 weeks and at 3 months
  The Global Assessment Scale for Children measures global functioning on a scale that ranges from 0 to 100 with higher scores indicating higher global functioning.
Brunnsviken Brief Quality of Life (BBQ) | Change from baseline at 7 weeks and at 3 months
  Brunnsviken Brief Quality of Life measures quality of Life in a total of 12 items (6 different areas of life). Satisfaction and how important the different areas of life are, are rated from 0-4. Total scores range from 0-96 with high scores indicating higher levels of quality of life.
Toronto Alexithymia Scale (TAS-20) | Change from baseline at 7 weeks and at 3 months
  Toronto Alexithymia Scale measures alexithymia. It contains a total of 20 items with 3 subscales (difficulties describing feelings: 7 items ranging from 7-35, difficulties identifying feelings: 5 items ranging from 5-25 and externally oriented thinking: 8 items ranging from 8-40). Total scores range from 20-100 with higher scores indicating higher levels of alexithymia.
Levels of Emotional Awareness (LEAS-C) | Change from baseline at 7 weeks and at 3 months
  Measures awareness of emotions, i.e., the ability to identify and describe own and others' emotions. The children's version used in the present study consists of 12 situations, in which the child is asked to describe which emotions he/she and another person would experience in a given situation. Answers are rated by an external rater on a five-grade scale divided into the three subscales: self, other and total.

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Zetterqvist, PhD, Principal Investigator — Region Ostergotland/Linköping universitet
Locations (1):
- Region Östergötland BUP-kliniken, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No